CLINICAL TRIAL: NCT06140589
Title: Study on the Efficacy, Safety and Cost-effectiveness of Cadonilimab in the Treatment of Cervical Cancer
Brief Title: Exploring the Efficacy, Safety and Cost-effectiveness Analysis of Cadonilimab in the Treatment of Cervical Cancer
Status: Recruiting | Type: Observational
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Fujian Medical University Affiliated Nanping First Hospital (Unknown); The First Hospital Affiliated to Fujian Medical University (Unknown); Fujian Medical University Union Hospital (Other); Gutian Hospital (Unknown); Jiangxi Provincial Cancer Hospital (Other); Shunde Women and Children's Hospital (Maternity and Child Healthcare Hospital of Shunde Foshan) (Unknown); Lianyungang Donghai County People&amp;amp;#39;s Hospital (Unknown); Changsha Maternal and Child Health Hospital (Unknown); Pingxiang Maternal and Child Health Hospital (Unknown); Huinan County People&amp;amp;#39;s Hospital (Unknown); People&amp;#39;s Hospital Affiliated to Fujian University of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: Sunyang1
Record Dates: First submitted 2023-11-06; First posted 2023-11-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; immune checkpoint inhibitors; Curative effect; safety; cost-effectiveness analysis
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- effective group: The tumor size of each diameter of the tumor before and after treatment was measured on magnetic resonance imaging or CT. According to Recist 1.1 criteria, patients who were evaluated as complete remission, partial remission and stable disease were included in the effective group. Patients assessed as having progressive disease were included in the treatment-refractory group.
  Interventions: Drug: Cadonilimab
- ineffective group: The tumor size of each diameter of the tumor before and after treatment was measured on magnetic resonance imaging or CT. According to Recist 1.1 criteria. Patients assessed as having progressive disease were included in the ineffective group.
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — The intravenous dose of Cadonilimab was 10mg/kg, and every 3 weeks was a course of treatment; Or 6mg/kg, every 2 weeks for a course of treatment

SUMMARY:
Cadonilimab, a PD-1/CTLA-4 bi-specific antibody, is being developed by Akeso, Inc. for the treatment of a range of solid tumors, including cervical cancer, lung cancer, gastric/gastroesophageal junction cancer, liver cancer and nasopharyngeal cancer. Cadonilimab was approved in China in June 2022 for use in patients with relapsed or metastatic cervical cancer who have progressed on or after platinum-based chemotherapy. The clinicopathological data of patients with persistent, recurrent or metastatic cervical cancer treated with Cadonilimab were collected, and medical images (magnetic resonance, CT, etc.) before and after treatment were followed up, and the efficacy was evaluated according to RECIST standards. The incidence and severity of adverse events and clinically significant abnormal laboratory test results were collected to evaluate the safety of the drug. Survival benefit analysis is conducted based on the patient's survival time and medical expenses.

DETAILED DESCRIPTION:
1. To explore the efficacy of Cadonilimab in the treatment of persistent, recurrent or metastatic cervical cancer.

   The size of each diameter of the tumor before and after treatment was measured on magnetic resonance imaging or CT. Complete response (CR) is defined as the complete disappearance of all target lesions. Partial response (PR): The sum of the diameters of all measurable target lesions is ≥30% below baseline. Disease progression (PD): The minimum value of the sum of the diameters of all measured target lesions during the entire experimental study is used as the reference, and the relative increase in the diameter sum is at least 20% (if the baseline measurement value is the smallest, the baseline value is used as the reference). Stable disease (SD): The reduction of the target lesion does not reach the PR level, and the increase does not reach the PD level, but is somewhere in between. For details, refer to the "Response Evaluation Criteria in Solid Tumors RECIST 1.1.
2. Observation on the safety and adverse reactions of Cadonilimab. Collect adverse events of tumors and abnormal laboratory indicators during medication (nausea, vomiting, bone marrow suppression, liver damage, rash, abnormal thyroid function, adrenocortical dysfunction, diabetes, myocarditis, myositis, hand-foot syndrome, etc.).
3. To explore the cost-benefit analysis of Cadonilimab in patients with cervical cancer.
4. Explore the relationship between genetic mutations and drug efficacy.

ELIGIBILITY:
Inclusion Criteria:

* •Persistent, recurrent or metastatic cervical cancer;

  * The pathological types are squamous cell carcinoma, adenocarcinoma, and adenosquamous carcinoma;
  * No combination with other multiple primary cancers;
  * MRI before treatment Or CT examination, according to RECIST evaluation standards, there is at least one measurable lesion;
  * ECOG score 0-1 points.
  * Subjects gave informed consent, voluntarily cooperated with clinical follow-up, and signed informed consent forms.

Exclusion Criteria:

* Patients with other histopathological types of cervical cancer, such as small cell carcinoma, clear cell carcinoma, sarcoma, etc.;

  * Previous treatment with immune checkpoint inhibitors;
  * There are drug contraindications, such as liver function Insufficiency, renal insufficiency, etc.
  * The patient withdraws the informed consent;
  * The researcher determines that the patient is not suitable to participate in this clinical study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic cervical cancer who were treated from June 2022 to December 2026 and met the above inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Cadonilimab in the treatment of persistent, recurrent or metastatic cervical cancer | 2026-12-21
  Objective response rate (ORR) was used to evaluate the efficacy of Cadonilimab in the treatment of advanced, recurrent or metastatic cervical cancer.
Efficacy of Cadonilimab in the treatment of persistent, recurrent or metastatic cervical cancer | 2026-12-21
  Progression free survival (PFS) was used to evaluate the efficacy of Cadonilimab in the treatment of advanced , recurrent or metastatic cervical cancer.
Efficacy of Cadonilimab in the treatment of persistent, recurrent or metastatic cervical cancer | 2026-12-21
  Disease control rate (DFS) was used to evaluate the efficacy of Cadonilimab in the treatment of advanced , recurrent or metastatic cervical cancer.
Efficacy of Cadonilimab in the treatment of persistent, recurrent or metastatic cervical cancer | 2026-12-21
  Overall survival (OS) was used to evaluate the efficacy of Cadonilimab in the treatment of advanced , recurrent or metastatic cervical cancer.

SECONDARY OUTCOMES:
Safety and adverse reactions of Cadonilimab | 2026-12-21
  According to CTCAE v5.0, any adverse events that occur to all subjects during the study period will be recorded. We recorded the clinical manifestation characteristics, severity, onset time, duration, treatment method and prognosis, and determined the correlation with Cadonilimab.
cost-effectiveness analysis of using Cadonilimab to treat cervical cancer | 2026-12-21
  The main economic outcome is the ICER.Health benefits were expressed as life years (LYs), and quality-adjusted life-years (QALYs) gained. The ICER was calculated by dividing the incremental cost difference between the two strategies, by the incremental difference in health outcomes (LYs and QALYs). Probabilistic Sensitivity Analysis (PSA) was performed to assess the impact of uncertainty around the key parameters of the model on the ICER. A second-order Monte Carlo simulation with 1000 iterations was used to run replicated outcomes. The normal distributions used for costs, utility and reimbursement ratio were carried to the specific limits.
The relationship between genetic mutations and the efficacy of Cadonilimab A in patients with cervical cancer | 2026-12-21
  According to the objective response rate, the patients in the study were divided into effective group and ineffective group. Whole exome sequencing was performed on some patients in the two groups to compare the differences in gene expression between the two group.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 420 Fuma Road, Jin'an District, Fuzhou City, Fujian Province, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
All relevant patient personal information and follow-up results of this study were saved by the principal investigator, and there was no plan to share them with other investigators

REFERENCES:
- [Background] Doroshow DB, Bhalla S, Beasley MB, Sholl LM, Kerr KM, Gnjatic S, Wistuba II, Rimm DL, Tsao MS, Hirsch FR. PD-L1 as a biomarker of response to immune-checkpoint inhibitors. Nat Rev Clin Oncol. 2021 Jun;18(6):345-362. doi: 10.1038/s41571-021-00473-5. Epub 2021 Feb 12. PMID 33580222
- [Background] Keam SJ. Cadonilimab: First Approval. Drugs. 2022 Aug;82(12):1333-1339. doi: 10.1007/s40265-022-01761-9. PMID 35986837
- [Background] Gao X, Xu N, Li Z, Shen L, Ji K, Zheng Z, Liu D, Lou H, Bai L, Liu T, Li Y, Li Y, Fan Q, Feng M, Zhong H, Huang Y, Lou G, Wang J, Lin X, Chen Y, An R, Li C, Zhou Q, Huang X, Guo Z, Wang S, Li G, Fei J, Zhu L, Zhu H, Li X, Li F, Liao S, Min Q, Tang L, Shan F, Gong J, Gao Y, Zhou J, Lu Z, Li X, Li J, Ren H, Liu X, Yang H, Li W, Song W, Wang ZM, Li B, Xia M, Wu X, Ji J. Safety and antitumour activity of cadonilimab, an anti-PD-1/CTLA-4 bispecific antibody, for patients with advanced solid tumours (COMPASSION-03): a multicentre, open-label, phase 1b/2 trial. Lancet Oncol. 2023 Oct;24(10):1134-1146. doi: 10.1016/S1470-2045(23)00411-4. PMID 37797632
- [Background] Frentzas S, Gan HK, Cosman R, Coward J, Tran B, Millward M, Zhou Y, Wang W, Xia D, Wang ZM, Li B, Xia M, Desai J. A phase 1a/1b first-in-human study (COMPASSION-01) evaluating cadonilimab in patients with advanced solid tumors. Cell Rep Med. 2023 Nov 21;4(11):101242. doi: 10.1016/j.xcrm.2023.101242. Epub 2023 Oct 17. PMID 37852261
- [Background] Zhang T, Lin Y, Gao Q. Bispecific antibodies targeting immunomodulatory checkpoints for cancer therapy. Cancer Biol Med. 2023 Mar 24;20(3):181-95. doi: 10.20892/j.issn.2095-3941.2023.0002. PMID 36971124
- [Derived] Chen J, Yu H, Lin Y, Hu D, Liu L, Fan R, Zou J, Zang L, Lin Y, Lin R, Chen D, Weng X, Shen F, Wang S, Zeng W, Tian Q, Yi Y, Chen Y, Miao J, Zhang B, Zou Y, Gao F, Lian R, Yang L, Sun Y. Real-world data of cadonilimab in recurrent or metastatic cervical cancer in China: a multicentric study. Front Immunol. 2025 Jul 14;16:1611696. doi: 10.3389/fimmu.2025.1611696. eCollection 2025. PMID 40726978